CLINICAL TRIAL: NCT05905640
Title: One-stop PrEP Care Pathway to Simplify PrEP Delivery in Kenya: The One-Stop PrEP Care Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other); Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Principal Investigator, Kenneth K Mugwanya, Assistant Professor: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00015873; R01MH129234-01A1 (NIH)
Record Dates: First submitted 2023-05-12; First posted 2023-06-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
Keywords: PrEP; HIV Prevention; PrEP adherence; Sexual behavior
MeSH Terms: conditions — HIV Infections; Sexual Behavior | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial of twelve public health clinics assigned 1:1 to implement either the intervention of One stop PrEP care pathway or usual clinic flow as control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm- Usual PrEP care pathway (No Intervention): At clinics that will serve as contemporaneous control clinics, eligible persons will receive PrEP according to the current client flow, which typically involves multiple room consultations. Quality improvement strategies will be promoted throughout the implementation period.
- Intervention Arm- One Stop PrEP care pathway (Other): In a one-stop arm, the number of client consultation rooms in the PrEP care pathway will be reduced to a single consultation room. All core PrEP services that include HIV testing, risk assessment, clinical review PrEP initiation, prescription, dispensing, and follow-up will be performed in a one-stop consultation with a single provider. Quality improvement strategies will be promoted throughout the implementation period.
  Interventions: Other: Method of PrEP delivery and consultation

INTERVENTIONS:
Other: Method of PrEP delivery and consultation — All core PrEP services that include HIV testing, risk assessment, clinical review PrEP initiation, prescription, dispensing, and follow-up will be performed in a one-stop consultation with a single provider.
  Arms: Intervention Arm- One Stop PrEP care pathway

SUMMARY:
The goal of this cluster randomized study is to understand if using a One stop PrEP delivery model can improve the efficiency of PrEP service delivery, reduce the cost of providing PrEP and allow continuation on PrEP. The investigators will evaluate data from men and women ≥15 years of age unknown to be living with HIV seeking PrEP services at public health facilities in western Kenya.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of one-stop PrEP services in 12 public health facilities in Kenya. The core implementation strategies to optimize one-stop PrEP care will include training of healthcare providers, technical assistance, joint clinic supervision with the county health officials, and abstraction of program data regarding PrEP initiations and continuations including characteristics of PrEP users for quality improvement. Within this large program, the study team will recruit a nested observational cohort to obtain detailed complementary individual clinical, behavioral, and mental health outcomes (including for clients who discontinue PrEP).

ELIGIBILITY:
Inclusion Criteria:

* ≥15 years of age
* Accessing PrEP services at implementing clinics.
* Eligible for PrEP per Kenya national guidelines

For in-depth and key delivery informant interviews

* Able and willing to provide consent
* Provides services at participating clinics (healthcare providers)
* Key policy maker

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation | Years 2-4 of the study, up to 36 months.
  PrEP initiation will be measured by client start of PrEP use documented on the ministry of health (MOH) tools. Data will be abstracted from MOH tools by project dedicated staff from up to 2400 persons newly initiating PrEP at the participating clinics.
PrEP continuation | up to 12 months of PrEP use.
  PrEP continuation will determined by clinic visit attendance and pharmacy PrEP refills records obtained by abstraction of MOH clinic records.
PrEP adherence | Years 2-4 of the study, up to 36 months.
  PrEP adherence will be measured objectively by quantification of drug levels in dried blood spots obtained at random subset visits from clients returning for PrEP refills.
Acceptability | Throughout the study period, up to 36 months
  Acceptability will be determined as the perception among clients, providers, and stakeholder that one-stop PrEP services is agreeable to them. Mixed methods assessments, including user and provider surveys and qualitative interviews with users and providers will be utilized to measure acceptability. The Proctors implementation framework will be utilized to organize outcomes and to understand acceptability of one-stop and quality improvement measures at the user, clinic, and provider level. Investigators will comprehensively triangulate all data sources to understand how system, provider, and client factors interact to influence adoption.
Adoption | Throughout the study period, up to 36 months
  Adoption will be determined as the proportion and characteristics of facilities adopting one-stop services. Mixed methods assessments, including provider surveys and qualitative interviews with users and providers will be utilized to measure adoption. The Proctors implementation framework will be utilized to organize outcomes and to understand adoption of one-stop and quality improvement measures at the clinic and provider level. Investigators will comprehensively triangulate all data sources to understand how system, provider, and client factors interact to influence adoption.
Fidelity | Throughout the study period, up to 36 months
  Fidelity will be defined as the degree to which one-stop pathway and quality improvement measures are implemented as planned. Checklists and technical assistant (TA) reports will be used to study how implementation of one-stop pathway and quality improvement measures are implemented per protocol at provider and clinic level. Investigators will comprehensively triangulate all data sources to understand how system, provider, and client factors interact to influence adoption.
Total client wait time and staff time spent on PrEP services | Throughout the study period, up to 36 months
  Efficiency will be defined as client wait time and staff time spent on PrEP services. Time will be done by observing at least 50 clinical visits per arm to assess wait time and staff time spent on counseling, HIV testing, clinical review, and PrEP provision
Satisfaction with services | Throughout the study period, up to 36 months
  Satisfaction will be defined ad fulfillment or happiness with one-stop service experience. Within the program we will use cross-sectional quantitative exit surveys administered to random clients at clinic to understand quality of care services and satisfaction with services.
Sustainability | up to 12 months after technical assistance support is scaled back
  Sustainability will be defined as the number of clinics using one-stop at 6, 12 months after technical assistance (TA). Checklists and technical assistant reports will be used to document implementation of one-stop after technical assistance support is scaled back
  The Proctors implementation framework will be used to organize implementation outcomes. Investigators will comprehensively triangulate all data sources to understand how system, provider, and client factors interact to influence continuation of PrEP.

SECONDARY OUTCOMES:
Incremental cost of one-stop PrEP services, including costs averted, and reduced client wait times. | up to 36 months.
  Micro-costing studies will be conducted during the implementation of one-stop PrEP delivery in intervention clinics as well as the current practice arm using activity-based approaches for costs incurred (start-up activities, clinic-wide training, recruitment, PrEP service delivery, including HIV testing, PrEP drugs, Sexually transmitted infection (STI) treatment, creatinine testing, and follow-up) and direct program costs averted (health costs saved by averting HIV infections, personnel costs averted as result of providing PrEP in one stop).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mugwanya, MBChB, MS, PhD, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute -KEMRI, Kisumu, Kenya